CLINICAL TRIAL: NCT04104880
Title: Anxiety and Depression In Patients With Obstructive Sleep Apnoea Before and After Continuous Positive Airway Pressure: the ADIPOSA Study
Brief Title: Anxiety and Depression In Patients With Obstructive Sleep Apnoea Before and After Continuous Positive Airway Pressure
Acronym: ADIPOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: University Hospital Virgen de las Nieves (Other)
Responsible Party: Principal Investigator, Almudena Carneiro Barrera, Teaching and research academic staff, Universidad de Granada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADIPOSA-19
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Uncontrolled before-and-after study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Continuous Positive Airway Pressure (CPAP) group (Experimental): Three-month CPAP use
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Adults previously diagnosed with obstructive sleep apnoea will receive a three-month CPAP intervention

SUMMARY:
Continuous positive airway pressure (CPAP) is the gold-standard treatment for obstructive sleep apnoea (OSA), the most common sleep-disordered breathing in the overall population. CPAP has shown to be effective in reducing apnoea-hypopnoea index (AHI) as well as other OSA polysomnographic outcomes. However, the effectiveness of this device on OSA daily functioning and mood disturbances outcomes still remains unclear. The ADIPOSA study is aimed at determining the effects of three-month CPAP use on anxiety-depression symptoms in patients with OSA. Participants will be adults previously diagnosed with OSA who will be allocated to a CPAP-treatment group. Outcomes will be measured at baseline and intervention end-point (three months) including daytime sleepiness, daily functioning and mood (anxiety and depression symptoms), AHI, other neurophysical and cardiorespiratory polysomnographic outcomes, and body weight. ADIPOSA may serve to establish the effectiveness of CPAP on daytime functioning and mood disturbances commonly found on patients with OSA and, in turn, on other OSA outcomes related to anxiety-depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Previous clinical diagnosis of mild/moderate/severe OSA (AHI > 5) by a healthcare professional
* Use of CPAP
* Motivation to participate in the study
* Willing to provide informed consent

Exclusion Criteria:

* Presence of any other primary sleep disorder
* Presence of any mental disorder (including depression, anxiety, and addiction to alcohol or other substances)
* Presence of any other severe organic disease, except for those comorbid to OSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Change in anxiety symptoms measured by State-Trait Anxiety Inventory (STAI) | Three months
  Changes in state anxiety and trait anxiety components measured by STAI questionnaire after three-month CPAP usage
Change in depression symptoms measured by Beck's Depression Inventory-Fast Screen (BDI-FS) | Three months
  Changes in depression symptoms measured by BDI-FS questionnaire after three-month CPAP usage

SECONDARY OUTCOMES:
Change in apnoea-hypopnoea index (AHI) from baseline to post-intervention | Three months
  Change in apnoea (airflow reduction greater than or equal to 90%) and hypopnoea (airflow reduction greater than or equal to 30%) episodes per hour of sleep, from baseline to post-intervention.
Change in oxygen desaturation index (ODI) from baseline to post-intervention. | Three months
  Change in the number of oxygen desaturations greater than or equal to 4%/h from baseline to post-intervention.
Change in excessive daytime sleepiness (EDS) from baseline to post-intervention | Three months
  Change in the difficulty in maintaining a desired level of wakefulness, measured by the Epworth sleepiness scale (ESS) from baseline to post-intervention. ESS is a 4-point scale (0 = no chance of dozing, 1 = slight chance of dozing, 2 = moderate chance of dozing, 3 = high chance of dozing) that measures the usual chances of dozing off or falling asleep while engaged in eight different activities. An ESS total score from 0 to 9 is considered to be normal while an ESS total score > 9 indicates high daytime sleepiness.
Change in body mass index (BMI) | Three months
  Change in body mass index from baseline to post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gualberto Buela-Casal, PhD, Study Director — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carneiro-Barrera A, Diaz-Roman A, Guillen-Riquelme A, Buela-Casal G. Weight loss and lifestyle interventions for obstructive sleep apnoea in adults: Systematic review and meta-analysis. Obes Rev. 2019 May;20(5):750-762. doi: 10.1111/obr.12824. Epub 2019 Jan 4. PMID 30609450
- [Background] Carneiro-Barrera A, Amaro-Gahete FJ, Diaz-Roman A, Guillen-Riquelme A, Jurado-Fasoli L, Saez-Roca G, Martin-Carrasco C, Ruiz JR, Buela-Casal G. Interdisciplinary Weight Loss and Lifestyle Intervention for Obstructive Sleep Apnoea in Adults: Rationale, Design and Methodology of the INTERAPNEA Study. Nutrients. 2019 Sep 15;11(9):2227. doi: 10.3390/nu11092227. PMID 31540168
- [Background] Sanchez AI, Martinez P, Miro E, Bardwell WA, Buela-Casal G. CPAP and behavioral therapies in patients with obstructive sleep apnea: effects on daytime sleepiness, mood, and cognitive function. Sleep Med Rev. 2009 Jun;13(3):223-33. doi: 10.1016/j.smrv.2008.07.002. Epub 2009 Feb 7. PMID 19201228
- [Background] Jurado-Gamez B, Guglielmi O, Gude F, Buela-Casal G. Effects of continuous positive airway pressure treatment on cognitive functions in patients with severe obstructive sleep apnoea. Neurologia. 2016 Jun;31(5):311-8. doi: 10.1016/j.nrl.2015.03.002. Epub 2015 May 11. English, Spanish. PMID 25976943